CLINICAL TRIAL: NCT03873168
Title: Post-Market Evaluation of HEMOBLAST™ Bellows Performance and Safety in Open Gynecological, Urological, ENT, Head and Neck, and Vascular Surgeries
Brief Title: Post-Market Evaluation of HEMOBLAST™ Bellows in Open Gynecological, Urological, ENT, Head, Neck, and Vascular Surgeries
Acronym: NOBLE-Open
Status: Terminated | Type: Observational
Why Stopped: Indication withdrawn
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ETC 2018-001
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hemostasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: HEMOBLAST™ Bellows — Surgeon has chosen to use HEMOBLAST™ Bellows as an adjunct to hemostasis when control of minimal, mild, or moderate bleeding by conventional procedures is ineffective or impractical in gynecological, urological, vascular, ENT and head and neck surgeries.

SUMMARY:
A prospective, multi-center, multi-national single arm study to evaluate the performance and safety of HEMOBLAST™ Bellows in open gynecological, urological, ENT and head and neck, and vascular surgery.

DETAILED DESCRIPTION:
A prospective, multi-center, multi-national single arm study conducted in Austria, France, and Germany to evaluate the performance and safety of HEMOBLAST™ Bellows in open gynecological, urological, ENT, head and neck, and vascular surgery. Up to 120 subjects will be enrolled at up to 10 sites, with a minimum of 8 subjects enrolled in each surgical specialty.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Patient is undergoing a non-emergent open gynecological, urological, ENT, head and neck, or vascular surgery
* Patient is willing and able to give prior written informed consent for investigation participation;
* Patient is 18 years of age or older.

Intra-operative Inclusion Criteria

* Patient has one or more target bleeding sites (TBS) for which control of bleeding by conventional procedures is ineffective or impractical.
* The TBS(s) has been treated with HEMOBLASTTM Bellows as per their instructions for use.

Exclusion Criteria:

* Patient is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding;
* Patient has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
* Patient has religious or other objections to porcine, bovine, or human components;
* Patient has any significant coagulation disorder;
* Patient has any other contraindications, warnings, precautions of the Approved Instruction For Use of HEMOBLAST™ Bellows preventing his/ her inclusion
* Patient is not appropriate for inclusion in the clinical trial, per the medical opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing open gynecological, urological, ENT and head and neck, and vascular procedures that meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Achievement of Hemostasis | Intraoperatively, expected within 3-10 minutes of application
  The proportion of subjects for which hemostasis was achieved after application of HEMOBLAST™ Bellows.

SECONDARY OUTCOMES:
Re-bleeding at Target Bleeding Site | Intraoperative, prior to surgical closure of the subject
  The rate of target bleeding site re-bleeding after hemostasis has been achieved with HEMOBLAST™ Bellows
Re-operation due to bleeding | Post-operatively, expected within 1-30 days of the surgical procedure
  The rate of re-operation due to post-operative bleeding/hemorrhage after treatment with HEMOBLAST™ Bellows

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vilz, MD, Principal Investigator — Unversity Hospital Bonn
Locations (9):
- Uniklinikum, Salzburg, Austria
- France (4):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - CHU Grenoble, Grenoble
  - Hopital Saint-Joseph, Paris
  - Clinique Rive Gauche, Toulouse
- Germany (4):
  - Universitatsklinikum Bonn, Bonn
  - Kliniken der Stadt Koln, Krankenhaus Merheim, Cologne
  - Agaplesion Markus krankenhaus, Frankfurt
  - St Franzikus-Hospital, Münster

IPD SHARING:
Plan to Share IPD: Undecided